CLINICAL TRIAL: NCT01686191
Title: Pharmacogenomics of Calcineurin Inhibitor Nephrotoxicity in Cardiac Transplantation
Brief Title: Genetic Predictors of Renal Dysfunction Following Heart Transplantation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Jewish Health (Other)
Responsible Party: Sponsor
Other Study IDs: 12-0869; 12GRNT12040211 (Other Grant/Funding Number: American Heart Association); UL1TR002535 (NIH); TL1TR002533 (NIH)
Record Dates: First submitted 2012-09-12; First posted 2012-09-17 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Heart Transplantation; Chronic Renal Insufficiency
Keywords: heart transplantation; chronic renal insufficiency; pharmacogenomics; cyclosporine; tacrolimus
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Buccal cell and blood sample for genomic DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac transplant recipients

SUMMARY:
Kidney disease is a common problem after heart transplantation. It may be caused by anti-rejection medications such as cyclosporine or tacrolimus. However, the reason why some people develop kidney problems after a heart transplant, but other people do not, is not fully known. This study plans to learn more about the relationship between a person's genetic make-up (DNA; deoxyribonucleic acid) and the risk of kidney problems after a heart transplant. The long-term goal of this research is to identify genetic variations that may help predict the development of kidney problems after heart transplantation.

ELIGIBILITY:
Inclusion Criteria:

* cardiac-only transplant
* 18 years of age or older at the time of cardiac transplant
* 1 year or more post-cardiac transplant
* treatment with cyclosporine or tacrolimus following transplant

Exclusion Criteria:

* combined organ transplant
* decisionally impaired
* unable to read or speak English
* unable or unwilling to provide written informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac transplant clinic
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Chronic renal dysfunction | year 2 post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Christina L Aquilante, Pharm.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States